CLINICAL TRIAL: NCT05211570
Title: A Phase 1/2 Study to Assess the Safety, Pharmacokinetics, and Efficacy of Daily Intravenous AB8939 in Patients With Relapsed/Refractory Acute Myeloid Leukemia
Brief Title: AB8939 in Patients With Relapsed/Refractory Acute Myeloid Leukemia
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AB Science (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AB18001; 2020-005122-28 (EudraCT Number)
Record Dates: First submitted 2022-01-12; First posted 2022-01-27 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Acute Myeloid Leukemia Refractory; Acute Myeloid Leukemia, in Relapse; Myelodysplastic Syndrome Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; GATA2 Deficiency | interventions — venetoclax

STUDY DESIGN:
Intervention Model Description: Open-label, multi-centre, non-randomized, 2-part study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- AB8939 (Experimental): AB8939 administered as a single agent
  Interventions: Drug: AB8939
- AB8939 plus Venetoclax (Experimental): AB8939 administered in combination with venetoclax
  Interventions: Drug: AB8939; Drug: Venetoclax

INTERVENTIONS:
Drug: AB8939 — Intravenous injection (from an initial dose of 0.9 mg/m²)
Drug: Venetoclax — the recommended starting dose for AML indication is 100 mg. Dose escalating regimen as per SmPC.
  Arms: AB8939 plus Venetoclax

SUMMARY:
The primary objective is to define the safety and tolerability of AB8939 in patients with AML by determining the dose-limiting toxicities, the maximum tolerated dose, and the recommended dose for dose expansion study.

DETAILED DESCRIPTION:
This is a Phase 1/2, open-label, multi-center, non-randomized, 2-part study in patients with refractory and relapsed AML and refractory myelodysplastic syndrome.

Study AB18001 has a multi-stage design. The first part is a dose escalation study that aims to determine the safety, tolerability and pharmacokinetic profiles of consecutive daily intravenous administration of AB8939 in patients with refractory or relapsed AML or patients with refractory myelodysplastic syndrome, and to determine the recommended dose for the second-stage dose expansion study. This dose expansion study aims to determine the schedule for a Phase 2 trial in patients with relapsed/refractory AML and to also provide an early efficacy assessment of AB8939.

ELIGIBILITY:
DOSE ESCALATION STUDY

Key Inclusion Criteria:

* Patients with documented diagnosis of acute myeloid leukemia (AML) based on the last version of the World Health Organization classification and eligible to second or third line of treatment.
* Patients with documented diagnosis of refractory melyodisplastic syndrome in second or third line of treatment, and with high risk at prognosis based on the IPSS-R scoring system.
* ECOG performance status ≤ 1
* Patients are able to understand, sign, and date the written informed consent form at screening visit prior to any protocol-specific procedures
* Patients are able and willing to comply with study procedures as per protocol, including bone marrow biopsies

Key Exclusion Criteria:

* Patients eligible to a standard of care
* Patients eligible to hematopoietic stem cell transplantation (HSCT) at the time of inclusion
* Patients diagnosed with acute promyelocytic leukemia (M3)
* Patients with clinically active CNS leukemia
* Patients with HSCT within 100 days prior to the first administration of AB8939
* Women who are lactating/breastfeeding or who plan to breastfeed while on study
* Women with a positive pregnancy test

Other protocol-defined inclusion/exclusion criteria may apply

EXPANSION COHORT STUDY

Key Inclusion Criteria:

* Patients with documented diagnosis of acute myeloid leukemia (AML) based on the last version of the World Health Organization classification and eligible to second or third line of treatment.
* ECOG performance status ≤ 2
* Patients are able to understand, sign, and date the written informed consent form at screening visit prior to any protocol-specific procedures
* Patients are able and willing to comply with study procedures as per protocol, including bone marrow biopsies

Key Exclusion Criteria:

* Patients eligible to a standard of care
* Patients eligible to hematopoietic stem cell transplantation (HSCT) at the time of inclusion
* Patients diagnosed with acute promyelocytic leukemia (M3)
* Patients with clinically active CNS leukemia
* Patients with HSCT within 100 days prior to the first administration of AB8939
* Women who are lactating/breastfeeding or who plan to breastfeed while on study
* Women with a positive pregnancy test

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Rate of dose limiting toxicity (DLT) | Up to 56 days
  Identification of the Maximal Tolerated Dose for different dosing schedules

SECONDARY OUTCOMES:
Objective Response Rate | Up to 56 days
  The proportion of patients who have a partial or complete response to therapy

CONTACTS AND LOCATIONS:
Overall Officials: Norbert Vey, MD, Principal Investigator — Institut Paoli Calmettes, Marseille, France; Nicholas Short, MD, Principal Investigator — MD Anderson Cancer Center, Houston, Texas
Locations (10):
- MD Anderson Cancer Center, Houston, Texas, United States
- Institut Paoli Calmettes, Marseille, France
- National and Kapodistrian University of Athens NKUA · Department of Hematology and Bone marrow Transplantation Unit, Athens, Greece
- Spain (7):
  - General University Hospital of Alicantet (Hospital General Universitario Dr. Balmis de Alicante), Alicante
  - Hospital San Pedro de Alcantara, Cáceres
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Quirónsalud, Madrid
  - MD Anderson Cancer Center Madrid, Madrid
  - Clínica Universidad de Navarra, Pamplona
  - Virgen del Rocío University Hospital (Hospital Universitario Virgen del Rocío), Seville

REFERENCES:
- [Background] Goubard A, Humbert M, Mansfield C, Hermine O, Dubreuil P, et al. In Vivo Assessment of the Next Generation Microtubule-Destabilizing Agent AB8939 in Patient-derived Xenograft Models of Acute Myeloid Leukemia. Blood (2019) 134 (Supplement_1): 5142. doi.org/10.1182/blood-2019-127143
- [Background] Goubard A, Humbert M, Mansfield C, Hermine O, Dubreuil P, et al. AB8939, a Microtubule-Destabilizing Agent with Potential to Overcome Multidrug Resistance, is Active Across the Range (M0-M7) of Acute Myeloid Leukemia Subtypes. Blood (2019) 134 (Supplement_1): 5154. doi.org/10.1182/blood-2019-127021
- [Background] Humbert M, Goubard A, Mansfield C, Hermine O, Dubreuil P, et al. Anticancer Activity of a Highly Potent Small Molecule Tubulin Polymerization Inhibitor, AB8939. Blood (2019) 134 (Supplement_1): 2075. doi.org/10.1182/blood-2019-122540